CLINICAL TRIAL: NCT01245153
Title: Phase 2B Study of Rectal Ballooning Training in Female Urinary Incontinence
Brief Title: Rectal Balloon Training in Female Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Natthiya Tantisiriwat, MD, Assist (hon), Chulalongkorn University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REHAB_201011
Record Dates: First submitted 2010-11-17; First posted 2010-11-22 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence, Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rectal Balloon Training (Experimental): Subjects in combined RBT and PFMT group are taught Foley catheter insertion technique. The catheter is inserted into the rectum until the lower end of the balloon is 1 cm inside from the anus. Then the balloon is blown with clean water. Subjects will contract pelvic floor muscle in standing position by contracting the pelvic floor muscle, hold and count 1 to 5, then relax and count 1 to 5. Subjects are instructed to do the exercise 15 times/set, 3 sets/day, every day for 6 weeks.
  Interventions: Other: Rectal Balloon Training
- Control group (Active Comparator): Patients receive Pelvic floor muscle training without inserting any kinds of equipment.
  Interventions: Other: Pelvic floor muscle training (PFMT)

INTERVENTIONS:
Other: Rectal Balloon Training — Subjects in combined RBT and PFMT group are taught for foley catheter insertion technique. The catheter is inserted into the rectum until the lower end of the balloon is 1 cm inside from the anus. Then the balloon is blown with clean water starting at 10 cc. Then the volume is progress to 15 cc in 3rd week and 20 cc in 5th week
  Arms: Rectal Balloon Training
Other: Pelvic floor muscle training (PFMT) — Standard pelvic floor muscle exercise (Pelvic floor muscle training;PFMT) is assigned for 6 weeks.
  Arms: Control group

SUMMARY:
Urinary incontinence (UI) is a common and worldwide problem.Although pelvic floor muscle training(PFMT) is the standard recommendation for conservative treatment but some patients had difficulty doing PFMT. They could not locate the pelvic floor muscles, and so could not perform the PFMT properly or increase intensity of the exercise. The authors hypothesized that rectal balloon training(RBT) may improve patients' pelvic floor recognition as well as it is another option of progressive strengthening of pelvic floor muscle. This study's aim is to combine RBT with PFMT using the water-filled balloons of Foley catheters

DETAILED DESCRIPTION:
This study's aim is to combine RBT with PFMT using the water-filled balloons of Foley catheters. The catheter would be inserted into the rectum and used as a tool to help the patient recognize the pelvic floor muscles. The advantages of Foley catheters are that they are cheap, safe for contacting the mucosa, easy for self-insertion, and can be reused. Furthermore, we can increase the load of exercise by increasing the amount of water pushing into the balloon, and can use that as a tool for progressive resistive exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 25 - 70 years
* Have urinary incontinence problem
* Follow command
* Informed consent

Exclusion Criteria:

* Previous surgical correction of UI
* Use medications for treating overactive bladder symptoms
* Impaired recent and/or recall memory
* Brain and/or Spinal cord lesion
* Untreated Urinary tract infection
* Anal lesion which contradicted for inserting instrument
* Prolapsed rectum
* Prolapsed uterus
* History of pelvic injury
* Pregnancy

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | Change from baseline in pelvic floor muscle strength at 6 weeks
  Pelvic floor muscle strength will be assessed by biofeedback and recorded in unit of mmHg.

SECONDARY OUTCOMES:
Clinical symptoms | At the first time then 6 weeks later
  Clinical symptoms are assessed from questionaire and one-hour pad test

CONTACTS AND LOCATIONS:
Overall Officials: Natthiya Tantisiriwat, Principal Investigator — King Chulalongkorn Memorial Hospital

REFERENCES:
- [Background] Bols EM, Berghmans BC, Hendriks EJ, de Bie RA, Melenhorst J, van Gemert WG, Baeten CG. A randomized physiotherapy trial in patients with fecal incontinence: design of the PhysioFIT-study. BMC Public Health. 2007 Dec 20;7:355. doi: 10.1186/1471-2458-7-355. PMID 18096041
- [Background] Whitehead WE, Burgio KL, Engel BT. Biofeedback treatment of fecal incontinence in geriatric patients. J Am Geriatr Soc. 1985 May;33(5):320-4. doi: 10.1111/j.1532-5415.1985.tb07130.x. PMID 3989196
- [Background] De Paepe H, Renson C, Van Laecke E, Raes A, Vande Walle J, Hoebeke P. Pelvic-floor therapy and toilet training in young children with dysfunctional voiding and obstipation. BJU Int. 2000 May;85(7):889-93. doi: 10.1046/j.1464-410x.2000.00664.x. PMID 10792172
- [Background] Dannecker C, Wolf V, Raab R, Hepp H, Anthuber C. EMG-biofeedback assisted pelvic floor muscle training is an effective therapy of stress urinary or mixed incontinence: a 7-year experience with 390 patients. Arch Gynecol Obstet. 2005 Dec;273(2):93-7. doi: 10.1007/s00404-005-0011-4. Epub 2005 Jul 6. PMID 16001201
- [Background] Cammu H, Van Nylen M. Pelvic floor exercises versus vaginal weight cones in genuine stress incontinence. Eur J Obstet Gynecol Reprod Biol. 1998 Mar;77(1):89-93. doi: 10.1016/s0301-2115(97)00237-6. PMID 9550207
- [Background] Bo K, Talseth T, Holme I. Single blind, randomised controlled trial of pelvic floor exercises, electrical stimulation, vaginal cones, and no treatment in management of genuine stress incontinence in women. BMJ. 1999 Feb 20;318(7182):487-93. doi: 10.1136/bmj.318.7182.487. PMID 10024253
- [Background] Dumoulin C, Hay-Smith J. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD005654. doi: 10.1002/14651858.CD005654.pub2. PMID 20091581
- [Background] Bunyavejchevin S. Risk factors of female urinary incontinence and overactive bladder in Thai postmenopausal women. J Med Assoc Thai. 2005 Sep;88 Suppl 4:S119-23. PMID 16623015
- [Background] Sakondhavat C, Choosuwan C, Kaewrudee S, Soontrapa S, Louanka K. Prevalence and risk factors of urinary incontinence in Khon Kaen menopausal women. J Med Assoc Thai. 2007 Dec;90(12):2553-8. PMID 18386703
- [Background] Panugthong P, Chulyamitporn T, Tanapat Y. Prevalence and risk factors of urinary incontinence in Thai menopausal women at Phramongkutklao Hospital. J Med Assoc Thai. 2005 Nov;88 Suppl 3:S25-30. PMID 16858941
- [Background] Manonai J, Poowapirom A, Kittipiboon S, Patrachai S, Udomsubpayakul U, Chittacharoen A. Female urinary incontinence: a cross-sectional study from a Thai rural area. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jun;17(4):321-5. doi: 10.1007/s00192-005-0002-9. Epub 2005 Sep 24. PMID 16184317
- [Background] Minassian VA, Drutz HP, Al-Badr A. Urinary incontinence as a worldwide problem. Int J Gynaecol Obstet. 2003 Sep;82(3):327-38. doi: 10.1016/s0020-7292(03)00220-0. PMID 14499979
- [Result] Sung MS, Hong JY, Choi YH, Baik SH, Yoon H. FES-biofeedback versus intensive pelvic floor muscle exercise for the prevention and treatment of genuine stress incontinence. J Korean Med Sci. 2000 Jun;15(3):303-8. doi: 10.3346/jkms.2000.15.3.303. PMID 10895973
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322